CLINICAL TRIAL: NCT04366141
Title: The Impact of a Barrier Enclosure on Endotracheal Intubation Duration and First Pass Attempt - A Randomized Controlled Trial
Brief Title: COVID-19 (Coronavirus Disease 2019) Intubation Barrier Box
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anthony Chau, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H20-01270
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
Keywords: Personal protective equipment; Barrier box
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This will be a prospective, open-label, randomized controlled trial in which patients will be randomly allocated to two study groups on a 1:1 basis into:
  1. COVID-19 barrier box Intervention group: Anesthesiologists will use a COVID barrier box during intubation.
  2. Control group: Anesthesiologists will not use a COVID barrier box during intubation. Standard intubation procedures will be followed for intubation.
  A block randomization strategy, using a computer-generated sequence of random numbers, will be used. Randomization will occur preoperatively if consented patients meet the eligibility criteria and provide informed consent.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 barrier box intervention group (Experimental): Attending anesthesiologists will use a COVID-19 barrier box for intubating the patient participants of this group.
  Interventions: Device: COVID-19 barrier box
- Control group (No Intervention): Attending anesthesiologists will use standard intubation procedures.

INTERVENTIONS:
Device: COVID-19 barrier box — Attending anesthesiologists will use a plastic proprietary barrier enclosure for intubating patients in the intervention group to protect spreading aerosolized droplets from patient to health care provider.
  Arms: COVID-19 barrier box intervention group

SUMMARY:
The trial will be done to determine the impact of a barrier enclosure, COVID (coronavirus disease -19) barrier box on endotracheal intubation attempts, and duration. This study will be a prospective, open-label, randomized controlled trial. A total of 100 patients scheduled for elective surgery will be randomly assigned in two groups (intervention group and control group). Participating attending anesthesiologists will intubate the intervention group patients with COVID barrier box and the control group patients without the box. The anesthesiologists and the intervention group patients will be surveyed about their perception after the surgery. The result of this study will help in decision making about using COVID barrier box to minimize the viral transmission from patients to healthcare workers during the pandemic.

DETAILED DESCRIPTION:
Purpose:

To assess the time to tracheal intubation (TTI) and first-pass success rate for attending anesthesiologists intubating with COVID-related modifications with or without the use of a COVID barrier box.

Hypothesis:

Using a COVID barrier box for tracheal intubation with COVID-related modifications for attending anesthesiologists would be prolonged compared to not using one.

Justification:

Tracheal intubation is a high-risk time point for attending anesthesiologists to contract COVID. This risk can be minimized by using a proprietary barrier enclosure, COVID barrier box covering a patient's head and neck during intubation. It is crucial to estimate the intubation time and first-pass success rate of using a COVID barrier box for introducing it to intubate critically ill COVID patients. The finding of this study can lead to a ground-breaking measure to minimize viral transmission to healthcare workers during the pandemic.

Objectives:

The primary objective of the study is to determine the TTI as measured by an observer. The secondary objectives are to assess the first-pass success rate, the total time of airway manipulation, as well as anesthesiologists' perception of intubation difficulty, and patients' satisfaction.

Research Design:

This study will be a prospective, open-label, randomized controlled trial. Consented eligible patients will be randomly allocated in a 1:1 ratio to intervention or control groups. A computer-generated sequence of random numbers will be used to randomize patients between groups. Consented eligible attending anesthesiologists will use COVID barrier box for intubating the intervention group but not for the control group. Each anesthesiologist will perform one practice intubation on manikins with the COVID barrier box before initiation of the study. The locally instituted COVID-related modifications will be in place during the practice intubation and intubations during surgery for both groups. A third party observer will monitor intubation time. All attending anesthesiologists and intervention group patients will undertake a post-survey.

Statistical Analysis:

A total of 100 patients with 50 in each group will be included in the study to ensure 99% power to detect a clinically significant TTI difference. Data distribution will be assessed using the Shapiro-Wilk and D'Agostino tests. Time outcomes will be analyzed using t-test or Mann-Whitney test. The first-pass success rate and categorical data about intubation difficulty and patient satisfaction will be analyzed using Fisher's Exact test.

ELIGIBILITY:
Patient Participant Inclusion Criteria:

1. Healthy American Society of Anesthesiologists (ASA) Classification 1 or 2 adults scheduled for elective surgery requiring orotracheal intubation
2. 18 years of age or older
3. COVID negative (As defined by negative COVID swab plus absence of screening symptoms as defined by: Fever, Cough, Shortness of breath or difficulty breathing, Chills, Repeated shaking with chills, Muscle pain, Headache, Sore throat, New loss of taste or smell)

Anesthesiologist Participant Inclusion Criteria:

1. Attending Anesthesiologist
2. Have performed at least 5 prior intubations using McGrath videolaryngoscopes
3. Have performed at least 5 prior endotracheal intubations with the locally instituted COVID-related modifications
4. Must not have more than one prior experience with using the COVID barrier box on real patients (Prior to the study start; not inclusive of intubations done in the context of this study)
5. Have performed at least one practice intubation on a manikin with the COVID barrier box prior to initiation of study

Patient Participant Exclusion Criteria:

1. Patient refusal, inability to consent or cooperate
2. Claustrophobia
3. Body habitus not allowing physical fit into COVID barrier box
4. History of documented difficult airway
5. Risk factors for difficult airway (Mallampati 3 or 4, thyromental distance less than 6 cm, interincisor distance less than 4 cm, upper lip bite test 2 or 3, body mass index (BMI) 30 or above, macroglossia, airway edema, blood in airway, cervical immobility, or any other concerning features deemed by attending anesthesiologist)
6. Risk factors for gastric aspiration
7. Allergy to rocuronium

Anesthesiologist Participant Exclusion Criteria:

1. Refusal to consent
2. Do not meet any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Time to tracheal intubation (TTI) | This will be measured at the time of intubation for an elective surgical patient. It will take approximately 5 minutes.
  TTI is the time from when the laryngoscope blade passes between the patient's lips until the first upstroke of the capnograph trace. TTI will be measured by a third party observer outside of the operating room.

SECONDARY OUTCOMES:
First pass success rate | This will be measured at the time of intubation for an elective surgical patient within 150 seconds of initiating the first attempt to intubate.
  A first pass success refers to successful insertion of the McGRATH™ videolaryngoscope or endotracheal tube by an anesthesiologist on the first-attempt without withdrawing from the mouth in no longer than 150 seconds.
Total time of airway manipulation | This will be measured at the time of intubation for an elective surgical patient. It will take approximately 5 minutes.
  This refers to the time from the face mask seal being lifted to the first upstroke of the capnograph trace.
Number of intubation attempts | This will be filled out as part of a questionnaire after intubation is completed. It will take approximately 10 minutes to complete the full questionnaire..
  Participant anesthesiologists will report the number of intubation attempts that were needed to achieve successful intubation.
Number of Operators needed for intubation | This will be filled out as part of a questionnaire after intubation is completed. It will take approximately 10 minutes to complete the full questionnaire..
  Participant anesthesiologists will report the number of operators needed to assist in successfully intubating the participant.
Number of alternative techniques used for intubation | This will be filled out as part of a questionnaire after intubation is completed. It will take approximately 10 minutes to complete the full questionnaire..
  Participant anesthesiologists will report the number of alternative techniques used for intubation (if any) i.e. repositioning of patient, change of materials (blade, endotracheal (ET) tube, addition of stylette), change in approach (nasotracheal vs orotracheal), use of another technique (Fibreoptic bronchoscopy, intubating laryngeal mask airway (LMA)
Cormack-Lehane Grade for the first attempt of intubation | This will be filled out as part of a questionnaire after intubation is completed. It will take approximately 10 minutes to complete the full questionnaire..
  Participant anesthesiologists will report the Cormack-Lehane Grade for the first attempt of intubation.
Lifting force applied on laryngoscope blade | This will be filled out as part of a questionnaire after intubation is completed. It will take approximately 10 minutes to complete the full questionnaire..
  Participant anesthesiologists will report if the lifting force applied on laryngoscope blade was normal or increased.
Laryngeal pressure application | This will be filled out as part of a questionnaire after intubation is completed. It will take approximately 10 minutes to complete the full questionnaire..
  Participant anesthesiologists will report if laryngeal pressure, such as Backward Upward Rightward Pressure (BURP) not inclusive of cricoid pressure was applied or not.
Vocal cord position | This will be filled out as part of a questionnaire after intubation is completed. It will take approximately 10 minutes to complete the full questionnaire..
  Participant anesthesiologists will report the vocal cord position (either abduction or adduction).
Anesthesiologist perception of intubation difficulty | This will be filled out as part of a questionnaire after intubation is completed. It will take approximately 10 minutes to complete the full questionnaire..
  Participant anesthesiologists will report the difficulty experienced during the intubation from a scale of 0 to 10 with 0 being without difficulty and 10 being maximum difficulty.
Anesthesiologist perception of contributors to difficulty in intubation, if any | This will be filled out as part of a questionnaire after intubation is completed. It will take approximately 10 minutes to complete the full questionnaire..
  Participant anesthesiologists will report any contributors to difficulties in intubation, or state "none", if no difficulties were experienced.
Patient acceptability of the COVID Barrier Box | This question will be asked as part of a short questionnaire administered to patients when they meet the Post Anesthesia Care Unit (PACU) discharge criteria (usually 2 to 5 hours after surgery). It will take about 10 minutes to complete.
  Patients from the intervention group will report the acceptability of COVID barrier box. They will be asked "How acceptable did you find the use of the COVID barrier box?" and respond on a five-point scale (acceptable, slightly acceptable, neutral, slightly unacceptable, unacceptable).
Patient comfort with the COVID Barrier Box | This question will be asked as part of a short questionnaire administered to patients when they meet the Post Anesthesia Care Unit (PACU) discharge criteria (usually 2 to 5 hours after surgery). It will take about 10 minutes to complete.
  Patients from the intervention group will report their level of comfort experienced with the use of the COVID barrier box. They will be asked "How comfortable did you find the use of the COVID barrier box?" and will respond on a five-point scale (comfortable, slightly comfortable, neither, slightly uncomfortable, uncomfortable).
Patient comments on the COVID Barrier Box | This question will be asked as part of a short questionnaire administered to patients when they meet the Post Anesthesia Care Unit (PACU) discharge criteria (usually 2 to 5 hours after surgery). It will take about 10 minutes to complete.
  Patients from the intervention group will report any comments that they have on the COVID barrier box.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Chau, MD, Principal Investigator — University of British Columbia
Locations (1):
- Providence Health Care, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tran K, Cimon K, Severn M, Pessoa-Silva CL, Conly J. Aerosol generating procedures and risk of transmission of acute respiratory infections to healthcare workers: a systematic review. PLoS One. 2012;7(4):e35797. doi: 10.1371/journal.pone.0035797. Epub 2012 Apr 26. PMID 22563403
- [Background] Canelli R, Connor CW, Gonzalez M, Nozari A, Ortega R. Barrier Enclosure during Endotracheal Intubation. N Engl J Med. 2020 May 14;382(20):1957-1958. doi: 10.1056/NEJMc2007589. Epub 2020 Apr 3. No abstract available. PMID 32243118
- [Background] Sakles JC, Mosier J, Patanwala AE, Dicken J. Learning curves for direct laryngoscopy and GlideScope(R) video laryngoscopy in an emergency medicine residency. West J Emerg Med. 2014 Nov;15(7):930-7. doi: 10.5811/westjem.2014.9.23691. Epub 2014 Oct 29. PMID 25493156
- [Background] Mohr S, Weigand MA, Hofer S, Martin E, Gries A, Walther A, Bernhard M. Developing the skill of laryngeal mask insertion: prospective single center study. Anaesthesist. 2013 Jun;62(6):447-52. doi: 10.1007/s00101-013-2185-7. Epub 2013 Jun 6. PMID 23736891
- [Background] Maharaj CH, O'Croinin D, Curley G, Harte BH, Laffey JG. A comparison of tracheal intubation using the Airtraq or the Macintosh laryngoscope in routine airway management: A randomised, controlled clinical trial. Anaesthesia. 2006 Nov;61(11):1093-9. doi: 10.1111/j.1365-2044.2006.04819.x. PMID 17042849
- [Background] Joshi R, Hypes CD, Greenberg J, Snyder L, Malo J, Bloom JW, Chopra H, Sakles JC, Mosier JM. Difficult Airway Characteristics Associated with First-Attempt Failure at Intubation Using Video Laryngoscopy in the Intensive Care Unit. Ann Am Thorac Soc. 2017 Mar;14(3):368-375. doi: 10.1513/AnnalsATS.201606-472OC. PMID 27983871
- [Background] Savoldelli GL, Schiffer E, Abegg C, Baeriswyl V, Clergue F, Waeber JL. Learning curves of the Glidescope, the McGrath and the Airtraq laryngoscopes: a manikin study. Eur J Anaesthesiol. 2009 Jul;26(7):554-8. doi: 10.1097/eja.0b013e3283269ff4. PMID 19522050
- [Background] Wallace CD, Foulds LT, McLeod GA, Younger RA, McGuire BE. A comparison of the ease of tracheal intubation using a McGrath MAC((R)) laryngoscope and a standard Macintosh laryngoscope. Anaesthesia. 2015 Nov;70(11):1281-5. doi: 10.1111/anae.13209. Epub 2015 Sep 4. PMID 26336853
- [Background] Nouruzi-Sedeh P, Schumann M, Groeben H. Laryngoscopy via Macintosh blade versus GlideScope: success rate and time for endotracheal intubation in untrained medical personnel. Anesthesiology. 2009 Jan;110(1):32-7. doi: 10.1097/ALN.0b013e318190b6a7. PMID 19104167
- [Background] Cook TM, El-Boghdadly K, McGuire B, McNarry AF, Patel A, Higgs A. Consensus guidelines for managing the airway in patients with COVID-19: Guidelines from the Difficult Airway Society, the Association of Anaesthetists the Intensive Care Society, the Faculty of Intensive Care Medicine and the Royal College of Anaesthetists. Anaesthesia. 2020 Jun;75(6):785-799. doi: 10.1111/anae.15054. Epub 2020 Apr 1. PMID 32221970
- [Background] Jones PM, Armstrong KP, Armstrong PM, Cherry RA, Harle CC, Hoogstra J, Turkstra TP. A comparison of glidescope videolaryngoscopy to direct laryngoscopy for nasotracheal intubation. Anesth Analg. 2008 Jul;107(1):144-8. doi: 10.1213/ane.0b013e31816d15c9. PMID 18635480
- [Background] Yao WL, Wan L, Xu H, Qian W, Wang XR, Tian YK, Zhang CH. A comparison of the McGrath(R) Series 5 videolaryngoscope and Macintosh laryngoscope for double-lumen tracheal tube placement in patients with a good glottic view at direct laryngoscopy. Anaesthesia. 2015 Jul;70(7):810-7. doi: 10.1111/anae.13040. Epub 2015 Feb 27. PMID 25721326
- [Background] CDC. Coronavirus Disease 2019 (COVID-19) - Symptoms [Internet]. Centers for Disease Control and Prevention. 2020 [cited 2020 Apr 20]. Available from: https://www.cdc.gov/coronavirus/2019-ncov/symptoms-testing/symptoms.html
- [Background] Chan A. Should we use an "aerosol box" for intubation? :11.
- [Derived] Jen TTH, Gusti V, Badh C, Mehta S, Denomme J, Lockhart S, Shams B, Klaibert B, Chau A. The impact of a barrier enclosure on time to tracheal intubation: a randomized controlled trial. Can J Anaesth. 2021 Sep;68(9):1358-1367. doi: 10.1007/s12630-021-02024-z. Epub 2021 May 10. PMID 33973161